CLINICAL TRIAL: NCT04172012
Title: Use of Probiotics to Reduce Infections and Death and Prevent Colonization With Extended-spectrum Beta-lactamase Producing Bacteria, Among Newborn Infants in Haydom and Surrounding Area, Tanzania, a Randomized Controlled Clinical Trial
Brief Title: Use of Probiotics to Reduce Infections, Death and ESBL Colonisation
Acronym: ProRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haydom Lutheran Hospital (Other)
Collaborators: University of Bergen (Other); Helse Stavanger HF (Other Government); UiT The Arctic University of Norway (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019/1025
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Neonatal Sepsis
Keywords: Tanzania; East Africa; Antimicrobial resistance; Probiotics; Extended Spectrum Beta-Lactamase Producing Bacteria
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Placebo-controlled double-blinded randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational product (probiotic) and placebo product have both been produced by the same manufacturer and is delivered in identical bottles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Active Comparator): Study subjects receive probiotic mixture for 4 weeks
  Interventions: Biological: Labinic (R) probiotic mixture
- Placebo (Placebo Comparator): Study subjects receive placebo mixture for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Labinic (R) probiotic mixture — Labinic (R) probiotic mixture containing Lactobacillus acidophilus and Bifidobacterium infantis and B. breve
  Arms: Probiotic
Other: Placebo — Placebo mixture
  Arms: Placebo

SUMMARY:
This study examines the effect of oral probiotic treatment to newborns on preventing hospitalizations, death and colonization with Extended-spectrum beta-lactamase-producing Gram negative bacteria. Half of the babies will receive 4 weeks treatment with an oral mixture of the probiotic Labinic (R) while the other half will receive a placebo mixture.

DETAILED DESCRIPTION:
Studies show that probiotics given to prematurely born babies prevents sepsis and is widely used in the western world for this purpose. Probiotics consists of one or more normal gut-bacteria. A large study in India showed that giving probiotics to full-born babies reduced hospitalizations and morbidity. This study investigates giving a probiotic mixture with different combination of bacteria, Lactobacillus acidophilus, Bifidobacterium infantis and Bifidobacterium breve, for a longer duration (4 weeks instead of 7 days).

Infections with antibiotic-resistant bacteria is a major threat to health-care world-wide, and sepsis/severe infection caused by such bacteria is a major cause of neonatal death. The study hypothesis is that giving probiotics to newborns prevents them from getting colonized with antibiotic-resistant bacteria, such as Extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL-PE). By preventing colonization with ESBL-PE, severe infections such as sepsis may be prevented, and thereby survival may be improved.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infants with a birth weight equal or above 2.0 kgs, will be included in the study between 0-3 days of life.
* Newborn infants have to come from families who are long-term or permanent residents in the defined catchment area for this trial (30 km radius from HLH) in Tanzania.
* Parents are able and willing to complete study visit (including required study procedures) schedules over the six months proposed follow-up, which also includes hospitalizations required for compliance of this study protocol.
* Parents agrees for the child not to participate in another study during the study period
* Children less than one year admitted to hospital with suspected infection, not included in the RCT, will be included in a sub-study. A separate inclusion form is prepared for these children.

Exclusion Criteria:

* Birth weight below 2 kg
* Other health problems/illness, obvious congenital malformations.
* Multiple pregnancy
* Parents not consenting

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Composite outcome hospitalization and death | 6 months from inclusion
  Primary outcome is hospitalization and/or death of study subject

SECONDARY OUTCOMES:
ESBL colonization | 6 weeks and 6 months
  Faecal colonisation with Extended-spectrum beta-lactamase-producing Enterobacteriaceae as detected by fecal swab
Hospitalisation | 6 weeks and 6 months
  Hospitalisation
Death | 6 months
  Death during study period
Body weight | 6 months
  Growth monitored by weight
Body length | 6 months
  Growth monitored by length
Stool microbiota | 6 weeks and 6 months
  Stool microbiota composition including resistome analysis (metagenome sequencing)
Stool metabolome | 6 weeks and 6 months
  Stool metabolome composition
Stool inflammatory markers - Calprotectin | 6 weeks and 6 months
  Levels of Calprotectin in participants' stool samples
Stool inflammatory markers - alpha-1 antitrypsin | 6 weeks and 6 months
  Levels of alpha-1 antitrypsin (AAT) in participants' stool samples
Stool inflammatory markers - myeloperoxidase | 6 weeks and 6 months
  Levels of human myeloperoxidase (MPO) in participants' stool samples
Number of participants with culture-confirmed bacteremia | 6 months
  Bacteremia confirmed by blood culture
Genetic characteristics of ESBL-producing Enterobacteriaceae | 6 weeks and 6 months
  Genetic characteristics of ESBL-E from colonization and clinical samples (targeted screening)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Langeland, MD, PhD, Principal Investigator — University of Bergen
Locations (1):
- Haydom Lutheran Hospital, Babati, Manyara Region, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panigrahi P, Parida S, Nanda NC, Satpathy R, Pradhan L, Chandel DS, Baccaglini L, Mohapatra A, Mohapatra SS, Misra PR, Chaudhry R, Chen HH, Johnson JA, Morris JG, Paneth N, Gewolb IH. A randomized synbiotic trial to prevent sepsis among infants in rural India. Nature. 2017 Aug 24;548(7668):407-412. doi: 10.1038/nature23480. Epub 2017 Aug 16. PMID 28813414
- [Background] Esaiassen E, Hjerde E, Cavanagh JP, Pedersen T, Andresen JH, Rettedal SI, Stoen R, Nakstad B, Willassen NP, Klingenberg C. Effects of Probiotic Supplementation on the Gut Microbiota and Antibiotic Resistome Development in Preterm Infants. Front Pediatr. 2018 Nov 16;6:347. doi: 10.3389/fped.2018.00347. eCollection 2018. PMID 30505830
- [Background] Tellevik MG, Blomberg B, Kommedal O, Maselle SY, Langeland N, Moyo SJ. High Prevalence of Faecal Carriage of ESBL-Producing Enterobacteriaceae among Children in Dar es Salaam, Tanzania. PLoS One. 2016 Dec 9;11(12):e0168024. doi: 10.1371/journal.pone.0168024. eCollection 2016. PMID 27936054
- [Derived] Moyo SJ, Justine M, Blomberg B, Lohr IH, Gideon J, Mdoe P, Mduma E, Manyahi J, Pettersen VK, Paschal J, Syre H, Bukhay R, Klingenberg C, Langeland N. Navigating the trials of a trial: lessons from ProRIDE on recruitment, retention, and follow-up in rural Africa. Trials. 2026 Jan 15. doi: 10.1186/s13063-026-09447-3. Online ahead of print. PMID 41535953
- [Derived] Klingenberg C, Justine M, Moyo SJ, Lohr IH, Gideon J, Mdoe P, Mduma E, Manyahi J, Bargheet A, Pettersen VK, Paschal J, Syre H, Bernhoff E, Bukhay R, Blomberg B, Langeland N. Home administration of a multistrain probiotic once per day for 4 weeks to newborn infants in Tanzania (ProRIDE): a double-blind, placebo-controlled randomised trial. Lancet Glob Health. 2025 Jun;13(6):e1082-e1090. doi: 10.1016/S2214-109X(25)00064-6. PMID 40412397
- [Derived] Kuwelker K, Langeland N, Lohr IH, Gidion J, Manyahi J, Moyo SJ, Blomberg B, Klingenberg C. Use of probiotics to reduce infections and death and prevent colonization with extended-spectrum beta-lactamase (ESBL)-producing bacteria among newborn infants in Tanzania (ProRIDE Trial): study protocol for a randomized controlled clinical trial. Trials. 2021 Apr 29;22(1):312. doi: 10.1186/s13063-021-05251-3. PMID 33926519

DOCUMENTS (3):
  • Study Protocol (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT04172012/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT04172012/SAP_001.pdf
  • Informed Consent Form (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT04172012/ICF_002.pdf